CLINICAL TRIAL: NCT04394468
Title: The Use of plasmaJet During Operative Laparoscopy for Endometriosis
Acronym: PLASMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2019/1742
Record Dates: First submitted 2020-02-10; First posted 2020-05-19 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient group (Other): Data is collected from women (18-45y) with endometriosis (superficial and / or deep infiltrating endometriosis) where the preferred treatment is a laparoscopic intervention at UZ Gent.
  Interventions: Device: PlasmaJet

INTERVENTIONS:
Device: PlasmaJet — Data will be collected during two contact moments, in particular during her admission for surgical laparoscopy, and during her postoperative check-up. Both of these are standard of care. No additional questionnaires will be taken. During the admission the postoperative pain scoreswill be monitored and collected. The duration of her stay in the hospital will also be recorded. During the postoperative check-up, which takes usually place six weeks after the surgery, complications will registered.

SUMMARY:
Endometriosis is a condition where functional endometrial tissue is present outside the uterus. It usually locates in the pelvis, which often includes the ovaries. One of the main concerns when performing surgery is to maintain fertility.

Nevertheless, a disadvantage of using monopolar and bipolar instruments for laparoscopic excision or coagulation of endometriosis lesions is the energy / thermal distribution that can cause damage to the surrounding healthy tissue. Therefore, the use of ultrasound, laser or plasma energy can potentially reduce damage to surrounding tissues and prevent adhesion formation. In addition, ablation of the internal surface of endometriomas can be an effective alternative to cystectomy.

The PlasmaJet system uses argon plasma which is released as kinetic, light and / or thermal energy. In this way the instrument can be applied within three functions, namely cutting, vaporizing and coagulating. Moreover, plasma will dissipate very quickly upon contact with tissue which consequently allows a controlled depth of tissue penetration. Thirdly, pure plasma energy differs from conventional electrosurgery since no electrical current will be spread through the tissue and therefore the thermal effect at surrounding tissues remains minimal.

The aim of this pilot study is to investigate the feasibility, effectiveness and safety of plasma energy in the treatment of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 45 years old.
* The presence of endometriosis; requiring surgical laparoscopy.

Exclusion Criteria:

* Women younger than 18 years.
* Women older than 45 years.
* Women who are scheduled for surgical laparoscopy where the removal of the uterus and / or ovaries is needed.
* Women who do not give written permission to participate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
feasibility of the PlasmaJet instrument | During laparoscopic surgery
  The surgeon's satisfaction with the use of plasma energy (5-point Likert scale).
effectiveness of the PlasmaJet instrument | During laparoscopic surgery
  - Whether or not to use additional instruments to achieve hemostasis (monopolar or bipolar coagulation) and / or complete resection of the lesions (monopolar or ultrasonic energy).
effectiveness of the PlasmaJet instrument | During laparoscopic surgery
  - completeness of resection or ablation, with a detailed description of deleted / ablated lesions.
effectiveness of the PlasmaJet instrument | During laparoscopic surgery
  - EFI score (Clinical instrument to predict pregnancy rates without IVF (ART) in patients after endometriosis surgery).
safety of the PlasmaJet instrument | During laparoscopic surgery until six weeks after surgery
  - Need for conversion to laparotomy.
safety of the PlasmaJet instrument | During laparoscopic surgery until six weeks after surgery
  - Serious complications up to 6 weeks after the operation. The most common complications that can occur with surgical laparoscopy are bleeding, damage to the surrounding tissues / structures and the formation of adhesions.
safety of the PlasmaJet instrument | During laparoscopic surgery until six weeks after surgery
  - Duration (in hours) of hospital stay after the procedure.
safety of the PlasmaJet instrument | During laparoscopic surgery until six weeks after surgery
  - Postoperative pain scores (VAS) (2 hours postoperatively, maximum pain scores during the days after surgery until the patient is discharged). Hereby the pain score is registered every hour during the stay in the PACU (Post-anesthesia care department). Afterwards, the pain score is recorded every four hours.

CONTACTS AND LOCATIONS:
Overall Officials: Tjalina Hamerlynck, Principal Investigator — University Hospital, Ghent
Locations (1):
- University hospital Ghent, Ghent, East-Flanders, Belgium